## **Informed Consent Form**

**Title of Study:** The Effect of a Physioterapy Program on the Emotional Well-being of Patiens Admitted to an Acute Hospitalization Unit

Principal Investigator: Sandra García Lobo

**Introduction:** You are invited to participate in a research study. Before you decide whether or not to participate, it is important that you understand why the research is being conducted and what it will involve. Please read the following information carefully and feel free to ask any questions you may have.

**Purpose of the Study**: The objective of this study is study the effectiveness of physiotherapy interventions on emotional well-being. By examining the impact of physiotherapy from a biopsychosocial perspective, this research aims to provide insights into the ways in which prolonged hospitalization affects patients' cognitive, social, and familial spheres. Moreover, it will highlight the necessity of integrating emotional support into physiotherapy practice.

**Procedures:** If you agree to participate in this study, you will recieve at least 4 physical terapeutic sessions in the unit where you are currently being hospitalized. The treatment will be adapted to the specific pathology, according to medical guidelines.

By participating in this clinical trial, you contribute to advancing medical research, potentially benefiting future patients with similar conditions. It is important to weigh these risks and benefits carefully. Please discuss any concerns or questions with your healthcare provider before consenting to participate in this trial. Confidentiality Your privacy is very important to us. All information collected during this study will be kept confidential. Your data will be coded and stored securely, and only authorized personnel will have access to it.

# **Voluntary Participation**

Your participation in this study is entirely voluntary. You may choose not to participate or to withdraw from the study at any time without any penalty or loss of benefits to which you are otherwise entitled.

### **Contact Information**

If you have any questions about this study, please contact:

Name: Sandra García Lobo

Telephone number: +34915202200 ext 19501

E-mail: sglobo@salud.madrid.org

### Consent

## **STATEMENTS AND SIGNATURES**

## PATIENT OR LEGAL GUARDIAN/RELATIVE

I have read and understood the information provided above. I have had the opportunity to ask questions, and all my questions have been answered to my satisfaction. I agree to participate in this study.

may withdraw my consent at any time

| As: PATIENT LEGAL GUARDIAN OR RELATIVE |
|----------------------------------------|
| Signed: |
| Date: |

## PRINCIPAL INVESTIGATOR

I have informed this participant and/or legal representative of the purpose and nature of the procedure described as well as its risks and alternatives.

| Signed: | · | |
|---------|---|------|
| Date: | | <br> |